CLINICAL TRIAL: NCT05644899
Title: Interlaminar Ultrasound-assisted or Landmark-based Intrathecal Administration of Nusinersen in Adult Patients With Spinal Muscular Atrophy: a Retrospective Analysis of More Than 500 Consecutive Administrations
Brief Title: Ultrasound-assisted or Landmark-based Intrathecal Administration of Nusinersen in Adult Patients With Spinal Muscular Atrophy (The EchoSpin Study)
Acronym: EchoSpin
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: EchoSpin
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2022-12

CONDITIONS: Anesthesia, Spinal; Spinal Puncture Complications; Spinal Muscular Atrophy; Ultrasonography
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SMA patients: 51 adults with a genetically confirmed diagnosis of SMA (13 SMA type 2, 38 SMA type 3) treated with nusinersen. The technique used was based on the anesthesiologist's preference.
  Interventions: Procedure: Interlaminar ultrasound-assisted intrathecal administration of nusinersen; Procedure: Landmark-based intrathecal administration of nusinersen

INTERVENTIONS:
Procedure: Interlaminar ultrasound-assisted intrathecal administration of nusinersen — All procedures were performed with patients either seated or placed in a lateral decubitus. After skin disinfection with 2% chlorhexidine in 70% alcohol, using a convex array, the L3-4 or L4-5 intervertebral space was identified and a left paramedian sagittal oblique view was obtained; the probe was rotated 90° into a transverse orientation, centered on the neuraxial midline, and moved in either the cephalad or caudal direction to obtain a transverse interlaminar view; the intersection between the two markings of the spinal midline and interspinous space was identified as the spinal entry point of the needle. After local anesthesia (LA) with lidocaine 2%, a 25-gauge non-traumatic 90 mm Whitacre spinal needle or a traumatic 90 mm Quincke spinal needle was used to access the subarachnoid space. After confirmation of cerebrospinal fluid (CSF) flow, 5 mL of CSF were removed. Subsequently, nusinersen was administered intrathecally over 1-3 min.
Procedure: Landmark-based intrathecal administration of nusinersen — All procedures were performed with patients placed in their most comfortable position (either seated or placed in a lateral decubitus). After skin disinfection with 2% chlorhexidine in 70% alcohol, conventional palpation of the superior aspect of iliac crest was performed and the palpated intercristal line was assumed to cross the spine at L4 vertebral body or L4-L5 interspace. The skin was marked with horizontal and vertical lines at the L3-L4 or L2-L3 interspaces and was referred as entry point of the needle. The procedure was then completed in the same fashion as for US-assisted technique.

SUMMARY:
Nusinersen (Spinraza, Biogen Inc, Boston, MA), the first treatment approved by FDA and EMA for all Spinal Muscular Atrophy (SMA) subtypes, is an antisense oligonucleotide that is administered intrathecally through a lumbar puncture. This procedure can be challenging in some adults with intermediate and late onset SMA (types II-IV) frequently presenting scoliosis secondary to neuromuscular weakness and often treated with spinal instrumentation to prevent worsening deformities.

In such patients, in order to access the intrathecal space, US guidance and/or assistance have been recently proposed as useful and successful tool. The US guidance and/or assistance have been associated to a high success rate, a reduction of number of attempts and needle passes to obtain a successful anesthesia. A reduced risk of adverse events (AEs), such as post dural puncture headache (PDPH) and low back pain (LBP), and low patient satisfaction often associated with multiple needle punctures was also reported.

Aim of this retrospective study was to report the efficacy, evaluated as rate of the successful procedures and subsequent delivery of nusinersen within the subarachnoid space, the number of attempts, the procedure time and the adverse events (AEs) of interlaminar intrathecal nusinersen administration using either ultrasound assistance or the landmark-based technique in a historical cohort of 51 adult SMA patients.

ELIGIBILITY:
Inclusion Criteria:

* A genetically confirmed diagnosis of SMA
* Treatment with nusinersen

Exclusion Criteria:

* congenital coagulopathy,
* localized infections,
* increased intracranial pressure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 51 adults with a genetically confirmed diagnosis of SMA (13 SMA type 2, 38 SMA type 3) consecutively treated with nusinersen intrathecal administration between April 2018 and August 2022 in "Policlinico A. Gemelli" in Rome.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Number of successful administrations | During the procedure
  Defined as a confirmation of the CSF flow through the spinal needle and subsequent administration of whole drug
Number of attempts | During the procedure
  Defined as the number of needle insertions through the skin surface
Procedure time | During the procedure
  The time in minutes from the start of US imaging or the palpation of superior aspect of iliac crest to visualization of CSF flow
Number of technical success procedures | During the procedure
  Defined as a successful intrathecal administration with equal or less than 4 attempts
Adverse events (AEs) | In the first 72 hours after the procedure
  Defined as mild AEs (Post Dural Puncture Headache, Low Back Pain) or severe AEs (spinal cord injury/epidural hematoma, abdominal organ lesions)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno A Zanfini, Principal Investigator — Fondazione Policlinico A. Gemelli
Locations (1):
- Fondazione Policlinico Gemelli, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No